CLINICAL TRIAL: NCT04894227
Title: A Double-blind, Randomized Clinical Trial to Evaluate the Lot-to-lot Consistency, Immunogenicity and Safety of an Inactivated SARS-CoV-2 Vaccine (CoronaVac） in Health Adults Aged 26-45 Years
Brief Title: Lot-to-lot Consistency of an Inactivated SARS-CoV-2 Vaccine for Prevention of COVID-19 in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-4001
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 inactivated vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inactivated SARS-CoV-2 vaccine Lot 1 (Experimental): Participants (n=360) aged 26-45 years will receive Inactivated SARS-CoV-2 vaccine Lot 1 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell）
- Inactivated SARS-CoV-2 vaccine Lot 2 (Experimental): Participants (n=360) aged 26-45 years will receive Inactivated SARS-CoV-2 vaccine Lot 2 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell）
- Inactivated SARS-CoV-2 vaccine Lot 3 (Experimental): Participants (n=360) aged 26-45 years will receive Inactivated SARS-CoV-2 vaccine Lot 3 according to 0,28-day immunization schedule.
  Interventions: Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell）

INTERVENTIONS:
Biological: Inactivated SARS-CoV-2 Vaccine (Vero cell） — 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac

SUMMARY:
This study is a double-blind, randomized phase Ⅳ clinical trial of the inactivated SARS-CoV-2 vaccine (CoronaVac）manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the lot-to-lot consistency, immunogenicity and safety of CoronaVac in healthy adults aged 26-45 years.

DETAILED DESCRIPTION:
This study is a double-blind, randomized phase Ⅳ clinical trial in healthy adults aged 26-45 years to evaluate the lot-to-lot consistency, immunogenicity and safety of the commercial-scale CoronaVac in healthy adults aged 26-45 years .The experimental vaccine was manufactured by Sinovac Research & Development Co.,Ltd. A total of 1080 healthy subjects aged 26 to 45 years old will be enrolled.The subjects will be randomly divided into three groups in a ratio of 1:1:1 to received two doses of vaccine on day 0 and day 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 26-45;
* The subjects can understand and voluntarily sign the informed consent form ;
* Proven legal identity.

Exclusion Criteria:

* Travel history / residence history of communities with case reports within 14 days prior to the study;
* History of contact with a SARS-CoV-2 infection (positive in nucleic acid test) within 14 days prior to the study;
* Have contacted patients with fever or respiratory symptoms from communities with case reports within 14 days prior to the study;
* Two or more cases of fever and / or respiratory symptoms in a small contact area of volunteers, such as home, office etc. within 14 days prior to the study;
* History of SARS-CoV-2 infection or receiving COVID-19 vaccine;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease (Systemic lupus erythematosus)or immunodeficiency / immunosuppression(HIV,history after organ transplantation)
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, spleenlessness, functional spleenlessness, spleenlessness or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months；
* Receipt of other investigational drugs in the past 30 days；
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Onset of various acute or chronic diseases within 7 days prior to the study;
* Axillary temperature >37.0°C;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 2 months;
* The subjects participated in other clinical trials during the follow-up period, or will be planned within 3 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 26 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1080 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer(GMT) of neutralizing antibody to live SARS-CoV-2 in susceptible population | Day 28 after the second dose
  GMT of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in susceptible population

SECONDARY OUTCOMES:
Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 in total population | Day 28 after the second dose
  Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in total population
Seropositivity rate of the neutralizing antibody to live SARS-CoV-2 in total population | Day 28 after the second dose
  Seropositivity rate of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in total population
GMT of the neutralizing antibody to live SARS-CoV-2 in total population | Day 28 after the second dose
  GMT of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in total population
Geometric mean increase (GMI) of the neutralizing antibody to live SARS-CoV-2 in total population | Day 28 after the second dose
  GMI of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in total population
Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 in susceptible population | Day 28 after the second dose
  Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in susceptible population
Seropositive rate of the neutralizing antibody to live SARS-CoV-2 in susceptible population | Day 28 after the second dose
  Seropositive rate of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in susceptible population
GMI of the neutralizing antibody to live SARS-CoV-2 in susceptible population | Day 28 after the second dose
  GMI of the neutralizing antibody to live SARS-CoV-2 at day 28 after the second dose in susceptible population
Seropositivity rate of anti-SARS-CoV-2 S antibody | Day 28 after the second dose
  Seropositivity rate of the anti-SARS-CoV-2 S antibody at day 28 after the second dose
Seroconversion rate of anti-SARS-CoV-2 S antibody | Day 28 after the second dose
  Seroconversion rate of the anti-SARS-CoV-2 S antibody at day 28 after the second dose
Geometric mean concentration (GMC) of anti-SARS-CoV-2 S antibody | Day 28 after the second dose
  GMC of the anti-SARS-CoV-2 S antibody at day 28 after the second dose
GMI of anti-SARS-CoV-2 S antibody | Day 28 after the second dose
  GMI of the anti-SARS-CoV-2 S antibody at day 28 after the second dose
Incidence of adverse reactions after vaccination | From the beginning of the vaccination to 28 days after the second dose
  Incidence of adverse reactions from the beginning of the vaccination to 28 days after the second dose

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Jingliang Wu, Huai'an, Jiangsu, China

REFERENCES:
- [Derived] Zhu D, Hu Y, Jiang Z, Yang T, Chu K, Zhang H, Hu J, Meng X, Tan Z, Wu J, Lian X, Li C, Pan H. Lot-to-lot consistency, immunogenicity, and safety of an inactivated SARS-CoV-2 vaccine (CoronaVac) in healthy adults: A randomized, double-blind, phase IV trial. Hum Vaccin Immunother. 2022 Nov 30;18(6):2135929. doi: 10.1080/21645515.2022.2135929. Epub 2022 Nov 28. PMID 36441137